CLINICAL TRIAL: NCT01287910
Title: Effect of Transmyocardial Laser Revascularization on Myocardial Perfusion and Left Ventricular Structure by Cardiovascular Magnetic Resonance Imaging and Dynamic Volumetric Computed Tomography
Brief Title: Transmyocardial Laser Revascularization and Cardiovascular Magnetic Resonance Imaging
Acronym: Amsterdam
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient population
Sponsor: Piedmont Healthcare (Other)
Collaborators: Cardiogenesis Corporation, a wholly-owned subsidiary of CryoLife, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Amsterdam
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-08

CONDITIONS: Angina; Chest Pain
Keywords: Cardiac; Angina; Chest pain
MeSH Terms: conditions — Angina Pectoris; Chest Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Patients (Other): All patients undergo the same study procedures
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — Cardiac MRI within 30 days prior to TMR procedure and 6 months after TMR procedure.

SUMMARY:
The primary goal of this study is to better understand how Transmyocardial Laser Revascularization (TMR) affects the functioning of the heart and, in turn, relieves angina in individuals with coronary heart disease using Magnetic Resonance (MR) images and Computed Tomography (CT) images in some patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or over
* Patients with medically refractory, severe, class III or IV angina based on the Canadian Cardiovascular Society angina scale as determined by a physician
* Ejection fraction 25% or greater
* Patients with significant ischemia in the myocardium and who are NOT candidates for treatment by direct coronary revascularization methods (i.e., CABG or PCI)
* Ability and willingness to consent and Authorization for use of PHI

Exclusion Criteria:

* Patient cannot undergo a surgical procedure or general anesthesia
* Patient not eligible for CMR study
* Severe unstable angina
* Q-wave MI within 3 weeks prior to TMR
* NQWMI within 2 weeks prior to TMR
* Decompensated heart failure (class III/IV) at the time of procedure
* Known increased bleeding risk
* Implanted pacemaker or defibrillator
* Clinically unstable arrhythmia
* Not able or willing to adhere to the study tests and procedures
* Inability or unwillingness to consent and Authorization for use of PHI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of coronary arteries with blood flow defects evaluated by magnetic resonance imaging (MRI) or computed tomography (CT) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Morris Brown, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States